CLINICAL TRIAL: NCT06833710
Title: Effect of Auricular Acupressure on Improving Sleep Quality in Nurses
Brief Title: Effect of Auricular Acupressure on Sleep Quality in Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Clinical trials office-Mackay Memorial Hospital, Mackay Memorial Hospital, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24MMHIS490e
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Auricular Acupressure 、Nurses、Sleep Quality
Keywords: Auricular Acupressure; Nurses; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Auricular Acupressure (Experimental): In the experimental group, the Shenmen point (MA-TF1) and Xin point (Xin MA) on both ears were treated with Wangbuliuxing seeds. Initially, the seeds were applied to the left ear for seven days, after which they were switched to the corresponding acupoints on the right ear. Following application, the seeds were pressed daily, once after each meal, with each acupoint being stimulated for 1 minute. The Chinese version of the Pittsburgh Sleep Quality Scale were measured on the day of application, as well as during the fourth and eighth weeks
  Interventions: Other: Auricular Acupressure

INTERVENTIONS:
Other: Auricular Acupressure — In the experimental group, the Shenmen point (MA-TF1) and Xin point (Xin MA) on both ears were treated with Wangbuliuxing seeds. Initially, the seeds were applied to the left ear for seven days, after which they were switched to the corresponding acupoints on the right ear. Following application, the seeds were pressed daily, once after each meal, with each acupoint being stimulated for 1 minute

SUMMARY:
The purpose of this study is to explore Effect of Auricular Acupressure on Improving Sleep Quality in Nurses. Adopting a quasi-experimental research design and convenience sampling, nursing staff from a northern medical center who scored 5 or higher on the Pittsburgh Sleep Quality Scale were selected as research subjects. Eligible participants were assigned to either the experimental group (auricular acupoint sticking) or the control group (no intervention).Pittsburgh Sleep Quality Scale were measured on the day of application, as well as during the fourth and eighth weeks. The collected data were analyzed using SPSS 29.0 for Windows.

DETAILED DESCRIPTION:
Background: Nursing staff face various pressures, shift systems, household responsibilities, and hormonal changes within the medical environment. They frequently experience issues such as sleep deprivation and inadequate rest, which can result in diminished work performance and increased fatigue. This, in turn, indirectly impacts the quality of care provided and heightens the risk to patient safety. Aim: Effect of Auricular Acupressure on Improving Sleep Quality in Nurses Methods: Adopting a quasi-experimental research design and convenience sampling, nursing staff from a northern medical center who scored 5 or higher on the Pittsburgh Sleep Quality Scale were selected as research subjects. Eligible participants were assigned to either the experimental group (auricular acupoint sticking) or the control group (no intervention). In the experimental group, the Shenmen point (MA-TF1) and Xin point (Xin MA) on both ears were treated with Wangbuliuxing seeds. Initially, the seeds were applied to the left ear for seven days, after which they were switched to the corresponding acupoints on the right ear. Following application, the seeds were pressed daily, once after each meal, with each acupoint being stimulated for 1 minute.Pittsburgh Sleep Quality Scale were measured on the day of application, as well as during the fourth and eighth weeks. The collected data were analyzed using SPSS 29.0 for Windows. Statistical analyses included percentages, means, chi-square tests, paired t-tests, independent t-tests, and generalized estimating equations to compare differences in sleep quality between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18
2. Nurses whose score on Pittsburgh Scale is greater than 5.
3. Those who are conscious, can communicate in Mandarin and Taiwanese, and answer the questionnaires in writing or orally, agree to participate in this study and sign the subject consent form.

Exclusion Criteria:

1. People with mental illness
2. infection or skin breakouts around the ears

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Scale | one year
  The Pittsburgh Sleep Quality Index includes seven factors: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan Presbyterian Church Mackay Medical Foundation Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No